CLINICAL TRIAL: NCT07084350
Title: Efficacy and Safety of Oral Lactulose Combined With Polyethylene Glycol Electrolytes Powder (PEG-ELS) for Bowel Preparation in Type II Diabetes Mellitus Patients: A Randomized Controlled Trial
Brief Title: Combination of Lactulose and Polyethylene Glycol Electrolytes Powder (PEG-ELS) for Bowel Preparation in Type II Diabetes Mellitus Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: XHNKKY-OLPG
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-06

CONDITIONS: Type II Diabetes Mellitus
Keywords: Type II diabetes mellitus; Bowel preparation; Lactulose; Polyethylene glycol
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Lactulose

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lac+PEG-ELS group (Experimental): Oral lactulose combined with PEG-ELS
  Interventions: Drug: lactulose; Drug: PEG (solution given 4 L)
- PEG-ELS group (Active Comparator): Only PEG-ELS
  Interventions: Drug: PEG (solution given 4 L)

INTERVENTIONS:
Drug: lactulose — 1. Two days before the colonoscopy: The patients should respectively take 30mL of lactulose orally on an empty stomach in the morning and at 8:00 PM of the same day, respectively.
  2. One Day Before the Colonoscopy: The patients should take 30mL of lactulose orally at 7:00 PM.
  3. On the Day of the Colonoscopy:
  For Morning Appointments:The patients should take 30mL of lactulose orally at 2:00 AM.
  For Afternoon Appointments:The patients should take 30mL of lactulose orally at 7:00 AM.
  Arms: Lac+PEG-ELS group
Drug: PEG (solution given 4 L) — 1. One Day Before the Colonoscopy: The patients should take 2000mL of PEG solution at 8:00 PM, and drink the entire solution within 2 hours.
  2. On the Day of the Colonoscopy:
  For Morning Appointments: The patients should take 2000mL of PEG solution at 3:00 AM and drink the entire solution within 2 hours.
  For Afternoon Appointments: The patients should take 2000mL of PEG solution at 7:00 AM and drink the entire solution within 2 hours.

SUMMARY:
Compared to the general population, diabetic patients have a significantly higher rate of inadequate bowel preparation. The European Society of Gastrointestinal Endoscopy (ESGE) guideline recommends polyethylene glycol (PEG) as the preferred bowel-cleansing agent, but there is currently no standardized bowel preparation protocol specifically for diabetic patients. Previous studies have shown that oral lactulose-based regimens or adding lactulose to the standard PEG protocol can improve bowel preparation quality, reduce adverse effects such as abdominal pain, bloating, nausea, and vomiting, and have no impact on blood glucose levels in diabetic patients after consuming 20g or 30g of lactulose. Herein, a multicenter randomized controlled trial(RCT) has been designed to explore the efficacy and safety of lactulose combined with polyethylene glycol electrolyte solution (PEG-ELS) for bowel preparation in patients with type II diabetes mellitus.

DETAILED DESCRIPTION:
Overall, 254 patients with type II diabetes mellitus will be enrolled. They will be randomly assigned at a ratio of 1:1 to the PEG group and lactulose +PEG group. The primary endpoint is the percentage of adequate bowel preparation. Secondary endpoints include the detection rates of polyps or adenomas and the incidence adverse reactions associated with bowel preparation (nausea, vomiting, abdominal pain, bloating, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. age 18~75 years;
2. patients undergoing colonoscopy;
3. diagnosis of type II diabetes mellitus；
4. sign the informed consent form.

Exclusion Criteria:

1. severe heart, lung or liver diseases;
2. bowel resection;
3. intestinal obstruction and massive ascites;
4. women preparing for pregnancy or those who were pregnant and lactating;
5. mental disorders;
6. dysphagia;
7. allergy to any medication used for bowel preparation;
8. have used prokinetic agents (such as domperidone or mosapride) within 14 days prior to the colonoscopy;
9. galactose or fructose intolerance, lactase deficiency, galactosemia, or glucose-galactose malabsorption syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
Adequate Bowel Preparation Rate | 3 days

SECONDARY OUTCOMES:
Adenoma and/or polyp detection rate (ADR/PDR) | 3 days
Adverse reactions rate associated with bowel preparation | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Background] American Diabetes Association Professional Practice Committee. 2. Diagnosis and Classification of Diabetes: Standards of Care in Diabetes-2025. Diabetes Care. 2025 Jan 1;48(1 Suppl 1):S27-S49. doi: 10.2337/dc25-S002. PMID 39651986
- [Background] Zhang X, Chen Y, Chen Y, Zhu W, Tang C, Lamm S, Li L. Polyethylene glycol combined with lactulose has better efficacy than polyethylene glycol alone in bowel preparation before colonoscopy: A meta-analysis. Clinics (Sao Paulo). 2023 Apr 3;78:100172. doi: 10.1016/j.clinsp.2023.100172. eCollection 2023. PMID 37019039
- [Background] He Y, Liu Q, Chen YW, Cui LJ, Cao K, Guo ZH. Bowel preparation protocol for hospitalized patients ages 50 years or older: A randomized controlled trial. World J Gastrointest Endosc. 2024 Jan 16;16(1):18-28. doi: 10.4253/wjge.v16.i1.18. PMID 38313462
- [Background] Yuanchao H, Xueping L, Tao L, Jianping N, Man M. The advantage of polyethylene glycol electrolyte solution combined with lactulose in patients with long interval preparation-to-colonoscopy. Turk J Gastroenterol. 2020 Jan;31(1):23-29. doi: 10.5152/tjg.2020.18888. PMID 32009610
- [Background] Ramos JA, Carvalho D, Arantes VN. Novel regimen for colonoscopy bowel preparation with oral lactulose: a prospective comparative study. Clin Endosc. 2024 Nov;57(6):775-782. doi: 10.5946/ce.2024.056. Epub 2024 Oct 22. PMID 39434557
- [Background] Li CX, Guo Y, Zhu YJ, Zhu JR, Xiao QS, Chen DF, Lan CH. Comparison of Polyethylene Glycol versus Lactulose Oral Solution for Bowel Preparation prior to Colonoscopy. Gastroenterol Res Pract. 2019 Apr 11;2019:2651450. doi: 10.1155/2019/2651450. eCollection 2019. PMID 31097959
- [Background] Lu J, Cao Q, Wang X, Pu J, Peng X. Application of Oral Lactulose in Combination With Polyethylene Glycol Electrolyte Powder for Colonoscopy Bowel Preparation in Patients With Constipation. Am J Ther. 2016 Jul-Aug;23(4):e1020-4. doi: 10.1097/MJT.0000000000000351. PMID 26658804
- [Background] Pieber TR, Svehlikova E, Mursic I, Esterl T, Wargenau M, Sartorius T, Pauly L, Schwejda-Guettes S, Neumann A, Faerber V, Stover JF, Gaigg B, Kuchinka-Koch A. Blood glucose response after oral lactulose intake in type 2 diabetic individuals. World J Diabetes. 2021 Jun 15;12(6):893-907. doi: 10.4239/wjd.v12.i6.893. PMID 34168736
- [Background] Chung YW, Han DS, Park KH, Kim KO, Park CH, Hahn T, Yoo KS, Park SH, Kim JH, Park CK. Patient factors predictive of inadequate bowel preparation using polyethylene glycol: a prospective study in Korea. J Clin Gastroenterol. 2009 May-Jun;43(5):448-52. doi: 10.1097/MCG.0b013e3181662442. PMID 18978506
- [Background] Hassan C, East J, Radaelli F, Spada C, Benamouzig R, Bisschops R, Bretthauer M, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Fuccio L, Awadie H, Gralnek I, Jover R, Kaminski MF, Pellise M, Triantafyllou K, Vanella G, Mangas-Sanjuan C, Frazzoni L, Van Hooft JE, Dumonceau JM. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Aug;51(8):775-794. doi: 10.1055/a-0959-0505. Epub 2019 Jul 11. PMID 31295746
- [Background] Hochberg I, Segol O, Shental R, Shimoni P, Eldor R. Antihyperglycemic therapy during colonoscopy preparation: A review and suggestions for practical recommendations. United European Gastroenterol J. 2019 Jul;7(6):735-740. doi: 10.1177/2050640619846365. Epub 2019 Apr 20. PMID 31316777
- [Background] Alvarez-Gonzalez MA, Flores-Le Roux JA, Seoane A, Pedro-Botet J, Carot L, Fernandez-Clotet A, Raga A, Pantaleon MA, Barranco L, Bory F, Lorenzo-Zuniga V. Efficacy of a multifactorial strategy for bowel preparation in diabetic patients undergoing colonoscopy: a randomized trial. Endoscopy. 2016 Nov;48(11):1003-1009. doi: 10.1055/s-0042-111320. Epub 2016 Aug 4. PMID 27490086
- [Background] Prasad VG, Abraham P. Management of chronic constipation in patients with diabetes mellitus. Indian J Gastroenterol. 2017 Jan;36(1):11-22. doi: 10.1007/s12664-016-0724-2. Epub 2016 Dec 17. PMID 27987136
- [Background] Chandrasekharan B, Anitha M, Blatt R, Shahnavaz N, Kooby D, Staley C, Mwangi S, Jones DP, Sitaraman SV, Srinivasan S. Colonic motor dysfunction in human diabetes is associated with enteric neuronal loss and increased oxidative stress. Neurogastroenterol Motil. 2011 Feb;23(2):131-8, e26. doi: 10.1111/j.1365-2982.2010.01611.x. Epub 2010 Oct 12. PMID 20939847
- [Background] Battle WM, Snape WJ Jr, Alavi A, Cohen S, Braunstein S. Colonic dysfunction in diabetes mellitus. Gastroenterology. 1980 Dec;79(6):1217-21. PMID 7439629
- [Background] Kim YH, Seo EH, Lee JS, Lee SH, Park HS, Choi SH, Park JY, Lee CW. Inadequate Bowel Cleansing Efficacy of Split-dose Polyethylene Glycol for Colonoscopy in Type 2 Diabetic Patients: A Prospective and Blinded Study. J Clin Gastroenterol. 2017 Mar;51(3):240-246. doi: 10.1097/MCG.0000000000000536. PMID 27136960
- [Background] Ozturk NA, Gokturk HS, Demir M, Unler GK, Gur G, Yilmaz U. Efficacy and safety of sodium phosphate for colon cleansing in type 2 diabetes mellitus. South Med J. 2010 Nov;103(11):1097-102. doi: 10.1097/SMJ.0b013e3181f20b13. PMID 20856180
- [Background] Amshoff Y, Maskarinec G, Shvetsov YB, Raquinio PH, Grandinetti A, Setiawan VW, Haiman CA, Le Marchand L. Type 2 diabetes and colorectal cancer survival: The multiethnic cohort. Int J Cancer. 2018 Jul 15;143(2):263-268. doi: 10.1002/ijc.31311. Epub 2018 Feb 25. PMID 29441528
- [Background] Yu GH, Li SF, Wei R, Jiang Z. Diabetes and Colorectal Cancer Risk: Clinical and Therapeutic Implications. J Diabetes Res. 2022 Mar 7;2022:1747326. doi: 10.1155/2022/1747326. eCollection 2022. PMID 35296101
- [Background] Wang M, Yang Y, Liao Z. Diabetes and cancer: Epidemiological and biological links. World J Diabetes. 2020 Jun 15;11(6):227-238. doi: 10.4239/wjd.v11.i6.227. PMID 32547697
- [Background] ASGE Standards of Practice Committee; Saltzman JR, Cash BD, Pasha SF, Early DS, Muthusamy VR, Khashab MA, Chathadi KV, Fanelli RD, Chandrasekhara V, Lightdale JR, Fonkalsrud L, Shergill AK, Hwang JH, Decker GA, Jue TL, Sharaf R, Fisher DA, Evans JA, Foley K, Shaukat A, Eloubeidi MA, Faulx AL, Wang A, Acosta RD. Bowel preparation before colonoscopy. Gastrointest Endosc. 2015 Apr;81(4):781-94. doi: 10.1016/j.gie.2014.09.048. Epub 2015 Jan 14. No abstract available. PMID 25595062
- [Background] Sharara AI, Abou Mrad RR. The modern bowel preparation in colonoscopy. Gastroenterol Clin North Am. 2013 Sep;42(3):577-98. doi: 10.1016/j.gtc.2013.05.010. PMID 23931861
- [Background] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Chan WK, Saravanan A, Manikam J, Goh KL, Mahadeva S. Appointment waiting times and education level influence the quality of bowel preparation in adult patients undergoing colonoscopy. BMC Gastroenterol. 2011 Jul 28;11:86. doi: 10.1186/1471-230X-11-86. PMID 21798022
- [Background] van Riswijk MLM, van Keulen KE, Siersema PD. Efficacy of ultra-low volume (</=1 L) bowel preparation fluids: Systematic review and meta-analysis. Dig Endosc. 2022 Jan;34(1):13-32. doi: 10.1111/den.14015. Epub 2021 Jun 24. PMID 33991373
- [Background] Wenqi S, Bei Z, Yunrong W, Xinrong W, Yifan L, Weiwei W, Muhan N, Peng Y, Xiaotan D, Wen L, Hua Y, Lei W, Min C. Lactulose vs Polyethylene Glycol for Bowel Preparation: A Single-Center, Prospective, Randomized Controlled Study Based on BMI. Clin Transl Gastroenterol. 2024 Jan 1;15(1):e00652. doi: 10.14309/ctg.0000000000000652. PMID 37795904